CLINICAL TRIAL: NCT05079282
Title: An Open-label, Multi-center, Non-randomized Phase I Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ONO-4685 Given as Monotherapy in Patients With Relapsed or Refractory T Cell Lymphoma
Brief Title: Study of ONO-4685 in Patients With Relapsed or Refractory T Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4685-03
Record Dates: First submitted 2021-09-30; First posted 2021-10-15 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Relapsed or Refractory T Cell Lymphoma
Keywords: ONO-4685; PD-1; CD3; Bispecific antibody; PTCL; AITL; PTCL-NOS; nodal PTCL with TFH; FTCL; CTCL; MF; SS
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ONO-4685 monotherapy (Experimental): Patients with relapsed or refractory T cell Lymphoma who meet eligibility criteria will be enrolled to receive ONO-4685 monotherapy
  Interventions: Drug: ONO-4685

INTERVENTIONS:
Drug: ONO-4685 — ONO-4685 is administered by IV infusion. The administration of ONO-4685 will be continued until disease progression or unacceptable toxicity is observed

SUMMARY:
This study will investigate the safety, tolerability, pharmacokinetics, and preliminary efficacy of ONO-4685 in patients with relapsed or refractory T cell Lymphoma

ELIGIBILITY:
Inclusion Criteria

1. Patients aged ≥ 18 years at time of screening
2. Written informed consent by the patient or the patients' legally authorized representative prior to screening
3. Patients with histologically or cytologically confirmed diagnosis of one of the following subtypes of T-cell lymphoma:

   1. Peripheral T-cell lymphoma (PTCL): Angioimmunoblastic T-cell lymphoma (AITL), PTCL, not otherwise specified (PTCL-NOS), nodal PTCL with T-follicular helper (TFH) and follicular T-cell lymphoma (FTCL)
   2. Cutaneous T-cell lymphoma (CTCL) (stages II-B, III, and IV): Mycosis fungoides (MF) and Sezary syndrome (SS)
4. Patients must have received at least 2 prior systemic therapies
5. Patients with PTCL must have at least 1 measurable lesion (Cheson BD, 2014)
6. Patients with CTCL must have assessable disease by response criteria for CTCL (Olsen EA, 2011)
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) = 0-2
8. Life expectancy of at least 3 months
9. Adequate bone marrow, renal and hepatic functions

Exclusion Criteria:

1. Patients with central nervous system (CNS) involvement
2. Patients with Adult T-cell leukemia/lymphoma (ATLL)
3. Prior allogeneic stem cell transplant
4. Prior treatment with ONO-4685, anti-PD-1, anti-PD-L1, anticytotoxic T lymphocyte associated protein 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
5. Prior allogeneic and autologous chimeric antigen receptor (CAR) T-cell therapy
6. Patients with malignancies (other than T-cell lymphoma) except for completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, or any other malignancies that has not relapsed for at least 2 years
7. History of severe allergy or hypersensitivity to any monoclonal antibodies, other therapeutic proteins or corticosteroid (e.g., dexamethasone)
8. History of infection with Mycobacterium tuberculosis within 2 years prior to the first dose of study treatment
9. Patients with systemic and active infection including human immunodeficiency virus (HIV), hepatitis B or C virus infection
10. Patients not recovered to Grade 1 or stabilized from the adverse effects (excluding alopecia) of any prior therapy for their malignancies
11. Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature, and severity of Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs). | Through study completion, an average of 1 year
  Adverse events with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 used as a guide for the grading of severity.
Estimate of Maximum Tolerate Dose (MTD) | Up to 3 weeks
  MTD will be estimated based on Dose limiting toxicity (DLT) observed during the first 3 weeks of treatment

SECONDARY OUTCOMES:
Plasma Concentration of ONO-4685 | Up to 48 weeks
  Plasma concentration will be assessed to evaluate Pharmacokinetics
Plasma Concentration of Anti-Drug Antibody (ADA) | Up to 48 weeks
  ADA to ONO-4685 will be assessed to evaluate potential immunogenicity.
Antitumor Activity of ONO-4685 | Through study completion, an average of 1 year
  Antitumor Activity of ONO-4685 will be assessed according to the response criteria for Lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of California Irvine Medical Center - Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - Yale Cancer Center, New Haven, Connecticut
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York-Presbyterian/Columbia University Irving Medical Center - Herbert Irving Comprehensive Cancer Center (HICCC), New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: No